CLINICAL TRIAL: NCT07345364
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single Ascending Doses of SIM0811 Injection in Healthy Chinese Adult Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIM0811-101
Record Dates: First submitted 2025-12-26; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Health, Subjective

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SIM0811 (Experimental): The study is designed to include 5 dose groups across 7 cohorts, with two administration methods: intravenous bolus plus intravenous infusion, and intravenous bolus alone. Each cohort will enroll 6 subjects to receive SIM0811 The study will employ a dose-escalation design starting from Cohort 1. After administration in each dose group/cohort, subjects will be observed for 7 days for safety evaluation. Provided no stopping criteria are met, escalation to the next dose level may proceed only after review by the Safety Review Committee (SRC)
  Interventions: Drug: SIM0811
- Placebo (Placebo Comparator): The study is designed to include 5 dose groups across 7 cohorts, with two administration methods: intravenous bolus plus intravenous infusion, and intravenous bolus alone. Each cohort will enroll 2 subjects to receive placebo The study will employ a dose-escalation design starting from Cohort 1. After administration in each dose group/cohort, subjects will be observed for 7 days for safety evaluation. Provided no stopping criteria are met, escalation to the next dose level may proceed only after review by the Safety Review Committee (SRC)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SIM0811 — The study will employ a dose-escalation design starting from Cohort 1. Each cohort will receive a single administration, sequentially completing Cohort 2, Cohort 3, Cohort 4, Cohort 5 , Cohort 6, and Cohort 7. After administration in each cohort, subjects will be observed for 7 days for safety evaluation. Provided no stopping criteria are met, escalation to the next dose level may proceed only after review by the Safety Review Committee (SRC).
  Arms: SIM0811
Drug: Placebo — The study will employ a dose-escalation design starting from Cohort 1. Each cohort will receive a single administration, sequentially completing Cohort 2, Cohort 3, Cohort 4, Cohort 5 , Cohort 6, and Cohort 7. After administration in each cohort, subjects will be observed for 7 days for safety evaluation. Provided no stopping criteria are met, escalation to the next dose level may proceed only after review by the Safety Review Committee (SRC).
  Arms: Placebo

SUMMARY:
This study plans to set up 5 dose groups across 7 cohorts, including intravenous bolus plus infusion administration as well as intravenous bolus alone. The study plans to enroll 8 subjects per cohort (investigational drug: placebo = 6:2), including both males and females, totaling 56 healthy subjects. The study begins with dose-escalation enrollment starting from Cohort 1. Each cohort receives a single dose, sequentially completing Cohorts 2, 3, 4, 5, 6, and 7. After each cohort's dosing is completed, a 7-day observation period is conducted for safety evaluation. If the termination criteria are not met, the study may proceed to the next dose level following assessment by the Safety Review Committee. By collecting adverse events, as well as abnormal indicators from vital signs, electrocardiograms, and laboratory tests, and collecting blood samples at planned time points to measure SIM0811 plasma concentration and thrombotic molecular markers, the study aims to evaluate the tolerability and safety of SIM0811 injection in Chinese healthy adult subjects, characterize its pharmacokinetic profile after single-dose administration, and explore the change curves of thrombotic molecular markers (plasmin-α2 antiplasmin complex PIC, fibrin degradation products FDP)

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Chinese male or female adults aged 18 to 45 years (inclusive), not pregnant and not breastfeeding.
2. Male subjects weight ≥50 kg, female subjects weight ≥45 kg, all ≤90 kg. Body Mass Index (BMI) between 19 and 26 kg/m² (inclusive). BMI = weight (kg) / height² (m²).
3. Female subjects must avoid the menstrual period during the trial. Subjects of childbearing potential must commit to no plan for pregnancy, sperm/egg donation within 2 weeks before screening and for 6 months after the last dose, and voluntarily adopt highly effective contraception (including partner).
4. Able to complete the study according to protocol requirements and commit to abstaining from smoking and alcohol during the trial.
5. Prior to the trial, have fully understood the nature, significance, potential benefits, possible inconveniences, and potential risks of the trial, voluntarily participate, can communicate well with the investigator, comply with all study requirements, and voluntarily sign the Ethics Committee-approved Informed Consent Form.

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded:

1. History of drug allergy, or specific allergies (asthma, urticaria, eczema, etc.), or allergic constitution (e.g., allergy to two or more drugs, foods, pollen), or known allergy or significant intolerance to the investigational product or any of its components.
2. Presence of clinically significant history of cardiovascular, respiratory, endocrine, urinary, digestive, hematological, neurological, skin, malignant tumor, infectious diseases, psychiatric disorders (e.g., seizures), metabolic abnormalities/dysfunction, etc.
3. Screening physical examination, vital signs, laboratory tests, or other examination results judged by the clinician as abnormal with clinical significance (confirmed upon repeat assessment); OR presence of the following abnormal laboratory indicators: Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), total bilirubin, direct bilirubin, creatinine above the upper limit of normal (ULN); platelet count below the lower limit of normal (LLN); hyperkalemia, hypokalemia, hypercalcemia, or hypocalcemia judged by the investigator as abnormal and clinically significant; PT prolongation > ULN + 3s, TT prolongation > ULN + 3s, APTT prolongation > ULN + 10s, INR > 1.2, FIB < 1.5 g/L or > 4.0 g/L, D-Dimer above ULN.
4. Screening ECG findings judged as abnormal with clinical significance. Resting heart rate not within the range of 50 to 100 beats per minute (exclusive of boundaries). QTcF interval > 470 ms (QTcF = QT/(RR)^0.33) or PR interval outside the range of 120 to 220 ms.
5. Risk factors for Torsades de Pointes, or family history (first-degree relatives - biological parents, siblings, or children) of short QT syndrome, long QT syndrome, unexplained sudden death at a young age (≤40 years), drowning, or sudden infant death syndrome.
6. Positive screening results for Hepatitis B surface antigen (HBsAg), Hepatitis C virus (HCV) antibody, Treponema pallidum specific antibody, or Human Immunodeficiency Virus (HIV) antibody.
7. Average daily alcohol consumption exceeding 2 units in the 2 years prior to screening, or weekly alcohol consumption >14 units (1 unit alcohol ≈ 360 ml beer or 45 ml 40% spirits or 150 ml wine); consumption of any alcohol-containing product within 24 hours prior to investigational product administration; or inability to stop alcohol consumption during the trial; or positive alcohol breath test.
8. Average daily cigarette consumption >5 in the 2 years prior to screening, or inability to stop using any tobacco products during the trial.
9. Positive screening result for drug abuse, or history of drug abuse or use of narcotics within the past five years.
10. Use of any prescription drugs, over-the-counter (OTC) drugs, Chinese herbal medicines, or health products within 2 weeks prior to screening and during screening, or within 5 half-lives of such drugs.
11. Any surgery or trauma within 1 year prior to investigational product administration that may affect trial safety or drug disposition, and judged by the investigator to be of current clinical significance; OR planned surgery during the trial or within 7 days after trial completion.
12. Difficulty with venous blood sampling, history of hematophobia or trypanophobia, or intolerance to indwelling venous catheter for blood sampling; OR history of phlebitis.
13. Blood donation or blood loss >200 ml within 3 months prior to screening, or receipt of blood transfusion or blood products within 4 weeks; OR plan to donate blood during the trial or within 3 months after trial completion.
14. History of blood abnormalities or related diseases, bleeding tendency, bleeding disorders (hemophilia, intracranial hemorrhage, gastrointestinal bleeding, urinary tract bleeding, hemoptysis, vitreous hemorrhage, etc.); OR arterial puncture at a site difficult to compress for hemostasis within 1 week prior; history of aneurysm.
15. Pregnancy, lactation, positive pregnancy test, sexual intercourse without protocol-required contraception within 2 weeks prior to screening, or planned pregnancy.
16. Vaccination within 1 month prior to screening, or planned vaccination during the trial / within 2 weeks after the last investigational product dose.
17. Participation in another drug or medical device clinical trial within 3 months prior to screening, or planned participation in another clinical trial during this study.
18. Special dietary requirements and unable to accept unified diet and schedule arrangements.
19. Other conditions judged by the clinical research physician as unsuitable for participation, or other reasons the subject may be unable to complete the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2026-01-13 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs), including type, incidence, grade (assessed according to NCI-CTCAE V5.0 criteria) | 7 days after final dose

SECONDARY OUTCOMES:
Peak plasma concentration(Cmax) of SIM0811 in serum | Within 1-2 weeks of final blood sample collection
Area Under the Concentration-time Curve from Time 0 to Time t of SIM0811 in serum | Within 1-2 weeks of final blood sample collection
Area Under the Concentration-time Curve from Time 0 to Infinity of SIM0811in serum | Within 1-2 weeks of final blood sample collection
Elimination Half-Life (T1/2) of SIM0811 in serum | Within 1-2 weeks of final blood sample collection

CONTACTS AND LOCATIONS:
Overall Officials: yuguo chen, Principal Investigator — Qilu Hospital of Shandong University; wei zhao, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No